CLINICAL TRIAL: NCT01652339
Title: Clinical Trial to Assess the Pharmacokinetic Characteristics of Lodivixx Tab. 5/160mg in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: HL-LDV-101
Record Dates: First submitted 2012-07-19; First posted 2012-07-30 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — Amlodipine, Valsartan Drug Combination; Amlodipine; Valsartan; levamlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exforge tab. 10/160mg (Active Comparator): * amlodipine besylate (10mg as amlodipine)
  * valsartan 160mg
  Interventions: Drug: Exforge tab. 10/160mg
- Lodivixx tab. 5/160mg (Experimental): * S-amlodipine nicotinate (5mg as S-amlodipine)
  * valsartan 160mg
  Interventions: Drug: Lodivixx tab. 5/160mg

INTERVENTIONS:
Drug: Exforge tab. 10/160mg
  Other Names: - amlodipine besylate; - valsartan
  Arms: Exforge tab. 10/160mg
Drug: Lodivixx tab. 5/160mg
  Other Names: - S-amlodipine; - valsartan
  Arms: Lodivixx tab. 5/160mg

SUMMARY:
To assess the pharmacokinetic characteristics of Lodivixx tab.5/160mg in healthy male subjects

* PK parameter evaluation
* Safety profile evaluation

ELIGIBILITY:
Inclusion Criteria:

* Years 20-45
* Body weight ≥ 50kg and 18 ≤ BMI ≤ 29kg/m2
* volunteer

Exclusion Criteria:

* Subject with serious active cardiovascular, respiratory, hepatologic, renal, hematologic, gastrointestinal, immunologic, dermal, neurologic, or psychological disease or history of such disease
* Subject with symptoms of acute disease within 28days prior to study medication dosing
* Subject with known for history which affect on the absorption, distribution, metabolism or excretion of drug
* Subject with clinically significant active chronic disease
* Subject with any of the following conditions in laboratory test i. AST(sGOT) or ALT(sGPT) > Upper normal limit × 1.5 ii. Total bilirubin > Upper normal limit × 1.5 iii. renal failure with Creatinine clearance < 50mL/min
* Clinically significant hypotension when screening period (SBP < 100mmHg, DBP < 60mmHg)
* Positive test results for HBs Ab, HCV Ab, Syphilis regain test
* Use of any prescription medication within 14 days prior to study medication dosing
* Use of any medication such as over-the-counter medication including oriental medication within 7 days prior to study medication dosing
* Subject with clinically significant allergic disease (except for mild allergic rhinitis and mild allergic dermatitis that are not needed to administer drug)
* Subject with known for hypersensitivity reaction to S-amlodipine, amlodipine and valsartan and dihydropyridine derivatives
* Subject who is not able to taking the institutional standard meal
* Subjects with whole blood donation within 60days, component blood donation within 20days
* Subjects receiving blood transfusion within 30days prior to study medication dosing
* Participation in any clinical investigation within 60days prior to study medication dosing
* Continued excessive use of caffeine (caffeine > five cups/day), alcohol(alcohol>30g/day) and severe heavy smoker (cigarette > 10 cigarettes per day)
* Subject who has been taken meal which affect on the absorption, distribution, metabolism, excretion of drug, especially grapefruit juice
* Subject taking inducer or inhibitor of drug metabolism enzyme such as barbital within 28days prior to study medication dosing
* Continued serum potassium concentration abnormal status (on baseline visit, < 3.5mEq/L or > 5.5mEq/L)
* Subjects with decision of nonparticipation through investigator's review due to laboratory test results or other excuse such as non-responding to request or instruction by investigator

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum concentration) | - Valsartan evaluation : 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48hr (14 points) - S-Amlodipine : 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 120, 168 (17 points)
AUC(area under curve) | - Valsartan evaluation : 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48hr (14 points) - S-Amlodipine : 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 120, 168 (17 points)

SECONDARY OUTCOMES:
Number of participants with adverse events | Participants will be followed for the duration of hospital stay, an expected average of 3 days and follow-up period for maximum 6 days from the discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jae Gook Shin, MD, Principal Investigator — Inje University
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea

REFERENCES:
- [Background] Plosker GL, Robinson DM. Amlodipine/Valsartan: fixed-dose combination in hypertension. Drugs. 2008;68(3):373-81. doi: 10.2165/00003495-200868030-00008. PMID 18257612